CLINICAL TRIAL: NCT04119219
Title: Collaborative Ocular Antiangiogenic Study of Ukraine. Multicentral, Open-label, Randomized, Prospective Study of Antiangiogenic Therapy of Choroidal Neovascularisation Associated With Angioid Streaks
Brief Title: Antiangiogenic Therapy of CNV Associated With Angioid Streaks
Acronym: COAST_UAasCNV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Filatov Institute of Eye Diseases and Tissue Therapy (Other)
Collaborators: Odessa National Medical University (Other); Mykolaiv Region Ophthalmogical Hospital (Other); Central Polyclinic of Internal Affairs of Ukraine (Other Government)
Responsible Party: Principal Investigator, Andrii Korol, MD, PhD, Head of Laser Department, The Filatov Institute of Eye Diseases and Tissue Therapy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0118U001612/3
Record Dates: First submitted 2019-10-07; First posted 2019-10-08 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Angioid Streaks of Macula
Keywords: fundus diseases; antiangiogenic therapy; subretinal neovascular membrane; intravitreal injection; anti-VEGF; angioid streaks
MeSH Terms: conditions — Angioid Streaks | interventions — Intravitreal Injections; Refractometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ranibizumab (Active Comparator): Arm 1
  Interventions: Procedure: Intravitreal injection
- Aflibercept (Active Comparator): Arm 2
  Interventions: Procedure: Intravitreal injection

INTERVENTIONS:
Procedure: Intravitreal injection — Intravitreal injection to the regimen pro re nata.
  Other Names: Patients after general ophthalmic examination (visometry, refractometry, biomicroscopy, ophthalmoscopy, OCT, fluorescent angiography) receive an injection according to the regimen pro re nata.

SUMMARY:
The purpose of this study is to determine the effectiveness of antiangiogenic therapy to choroidal neovascularization secondary to angioid streaks.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effectiveness of antiangiogenic therapy to choroidal neovascularization secondary to angioid streaks.

This study is planned as a follow-up. Patients with angioid streaks included in it will receive antiangiogenic therapy in accordance with the approved indications for use indicated in the instructions for the use of drugs in Ukraine.

The treatment proposed in this study is based on the world experience and scientific developments of the Filatov Institute of Eye Diseases and Tissue Therapy of the NAMS of Ukraine ". Therefore, it is expected that the benefit / risk ratio in relation to the participation in this study should not be different from that described in the scientific literature and the benefits outweigh the risk. It is known that the absence of treatment in these diseases leads to an irreparable loss of central vision.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

  1. Able to read (or, if unable to read due to visual impairment, be read to verbatim by the person administering the informed consent form or a family member) and understand the informed consent form and willing to sign the informed consent form.
  2. Signed informed consent form.
  3. Men and women ≥ 18 years of age.
  4. Willing, committed, and able to return for all clinic visits and complete all study-related procedures.
  5. First diagnosed active subfoveal or juxtafoveal (within 1 to 199 μm of the center of the fovea) CNV secondary to angioid streaks as defined by leakage on FA
  6. Transparent optical media and possibility to mydriasis.
  7. Best corrected visual acuity at least 20/100 Equivalent of Snellen (ETDRS).
* Exclusion Criteria:

  1. Ocular media of insufficient quality to obtain fundus and OCT images in the study eye.
  2. Recurrent CNV in the study eye.
  3. History or presence of CNV with an origin other than angioid streaks in the study eye.
  4. Ocular inflammation or external ocular inflammation in the study eye. 5 Concurrent disease in the study eye that would compromise BCVA or require medical or surgical intervention during the study period.

  6. Any ocular disorder in the study eye that, in the opinion of the investigator, may confound interpretation of the study results.

  7. Significant scarring or atrophy in the fovea that indicates substantial irreversible vision loss in the study eye.

  8. Evidence at examination of infectious blepharitis, keratitis, scleritis, or conjunctivitis in either eye or current treatment for serious systemic infection.

  9. Vitreomacular traction or traction retinal detachment, epiretinal membrane in either eye.

  10. Any iris neovascularization and/or vitreous hemorrhage in either eye. 11. Uncontrolled glaucoma, or previous filtration surgery in either eye. 12. Any prior or concomitant treatment with another investigational agent for CNV in the study eye.

  13. Any previous panretinal photocoagulation or subfoveal thermal laser therapy in the study eye.

  14. Any prior treatment with photodynamic therapy in the study eye. 15. Cataract surgery within 3 months prior to Day 1 in the study eye. 16. Yttrium-aluminum-garnet laser capsulotomy within 2 months prior to Day 1 in the study eye.

  17. Any other intraocular surgery within 3 months prior to Day 1 in the study eye.

  18. History of vitreoretinal surgery and/or scleral buckle surgery in the study eye.

  19. Any prior treatment with anti-VEGF agents. 20. Previous use of intraocular or periocular corticosteroids in either eye within 3 months prior to Day 1.

  21. Previous assignment to treatment during this study. 22. Uncontrolled hypertension. 23. History of cerebrovascular disease or myocardial infarction within 6 months prior to Baseline/Day 1.

  24. History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, may affect interpretation of the results of the study, or renders the subject at high risk from treatment complications.

  25. Women of childbearing potential without contraception, women who intend to breastfeed during the study. All subjects (both men and women) of childbearing potential who are unwilling to use adequate birth control measures during the course of the study.

  26. Renal failure requiring dialysis or renal transplant. 27. Participation in an investigational study within 30 days prior to Screening/Visit 1 that involved treatment with any drug (excluding vitamins and minerals) or device.

  28. Known serious allergy to the fluorescein sodium for injection in angiography or Verteporfin.

  29. Inability to obtain fundus photographs or fluorescein angiograms of sufficient quality

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-03-27 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Mean Change in Best Corrected Visual Acuity (BCVA) as Measured by ETDRS Chart | Baseline-Month 12
  Defined study baseline range of ETDRS equivalent of 20/200 to 20/20) in the study eye; a higher score represents better functioning.

SECONDARY OUTCOMES:
Mean Change in Central Retinal Thickness (CRT) as Assessed by Optical Coherence Tomography (OCT) | Baseline-Month 12
  A negative number indicates improvement (reduced thickness).
Average Number of Intravitreal Injections | Baseline-Month 12
  The number of intravitreal injections administered
Number of Endophthalmitis after Intravitreal Injections | Baseline-Month 12
  The number of endophthalmitis registered in patients after intravitreal injections

CONTACTS AND LOCATIONS:
Overall Officials: Andrii MD Korol, PhD, Principal Investigator — The Filatov Institute of Eye Diseases and Tissue Therapy
Locations (3):
- Ukraine (3):
  - Mykolaiv Region Ophthalmogical Hospital, Mykolaiv
  - Odessa National Medical University, Odesa
  - The Filatov Institute of Eye Diseases and Tissue Therapy, Odesa

IPD SHARING:
Plan to Share IPD: No